CLINICAL TRIAL: NCT02382120
Title: Accuracy and Precision of Non-invasive Effective Pulmonary Perfusion Measurement Using Volumetric Capnography
Brief Title: Accuracy of Non-invasive Effective Pulmonary Perfusion Measurement by CO2
Status: Completed | Type: Observational
Sponsor: Hospital Privado de Comunidad de Mar del Plata (Other)
Responsible Party: Sponsor
Other Study IDs: 23022015
Record Dates: First submitted 2015-03-03; First posted 2015-03-06 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-05

CONDITIONS: Cardiovascular Disease
Keywords: carbon dioxide; cardiac output; ventilation; thermodilution
MeSH Terms: conditions — Cardiovascular Diseases; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients undergoing cardiovascular surgery: Patients ASA 3-4 undergoing cardiac surgery.

SUMMARY:
Cardiac output monitoring is mandatory in most surgical and critical care patients. Many techniques to assess cardiac output are invasive and/or have many limitations, contraindications and drawbacks. The measurement of cardiac output throughout the CO2 signal is an interesting option due to the simplicity and non-invasive nature of its calculation.

The present study was designed to compare the cardiac output measurement using a capnodynamic formula versus the reference thermodilution method.

DETAILED DESCRIPTION:
This is a prospective and observational study designed to test the accuracy and precision of the non-invasive capnodynamic cardiac output measurement in mechanically ventilated patients. We will study 30 patients undergoing cardiovascular by pass in which an invasive trans-thoracic thermodilution method (PICCOScience) is indicated - the reference method.

A pair of thermodilutions and capnodynamic cardiac output measurement will be performed along the surgery. Analysis of precision will be done at the begining of the protocol and during stable hemodynamic conditions. Accuracy will then assessed using the Bland-Altmann plot and regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Programmed cardiac surgeries
* Surgeries with cardiopulmonary bypass

Exclusion Criteria:

* Emergency surgeries.
* Acute pulmonary diseases
* Contraindication of femoral catheters.
* Need of counter-pulsation baloon

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac surgical ASA II-III patients.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2018-04-21 (Actual); Study Completion 2018-07-21 (Actual)

PRIMARY OUTCOMES:
Accuracy and precision of capnodynamic to measure cardiac output | 8 months
  Comparison between a reference method (thermodilution) with a new one (capnodynamics)

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Tusman, MD, Principal Investigator — Hospital Privado de Comunidad de Mar del Plata
Locations (1):
- Hospital Privado de Comunidad, Mar del Plata, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Capek JM, Roy RJ. Noninvasive measurement of cardiac output using partial CO2 rebreathing. IEEE Trans Biomed Eng. 1988 Sep;35(9):653-61. doi: 10.1109/10.7266. No abstract available. PMID 3139547
- [Result] Peyton PJ, Venkatesan Y, Hood SG, Junor P, May C. Noninvasive, automated and continuous cardiac output monitoring by pulmonary capnodynamics: breath-by-breath comparison with ultrasonic flow probe. Anesthesiology. 2006 Jul;105(1):72-80. doi: 10.1097/00000542-200607000-00015. PMID 16809997